CLINICAL TRIAL: NCT03788850
Title: Factors Associated With Residual Disease In The Central Cone: A Disease Prediction Model
Brief Title: Factors Associated With Residual Disease In The Central Cone
Acronym: FARDCC
Status: Completed | Type: Observational
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, David Cantu, Chief of clinical trial departament, National Institute of Cancerología
Other Study IDs: 12102018INC
Record Dates: First submitted 2018-11-05; First posted 2018-12-28 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: residual disease; central cone; predictive model
MeSH Terms: conditions — Uterine Cervical Dysplasia; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cervical conization using the loop electrosurgical excision procedure (LEEP) is the standard treatment for patients with high-grade cervical intraepithelial neoplasia. Several studies have shown that excising a central cone reduces the rate of positive endocervical margins. The purpose of this study is to identify clinicopathological factors associated with residual disease in the central cone and to develop a predictive model to better determine which patients may require this additional procedure.

DETAILED DESCRIPTION:
This study pretends to create a retrospective database including all patient who underwent a loop electrosurgical excision procedure by treatment for high-grade cervical intraepithelial neoplasia and create a a predictive model for top-hat resection in patients with high grade CIN

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent a loop electrosurgical excision procedure (LEEP)

Exclusion Criteria:

* a diagnosis of micro-invasion or nonsquamous histology
* less than six months of follow-up
* incomplete information in their clinical charts.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent a cervical cone procedure at the Dysplasia Clinic of the Instituto Nacional de Cancerologia in Mexico City
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Identify the clinical and pathologic factors associated with residual disease | 1month
  Whit the variables identified as factors associated with the residual disease develop a predictive model to determine which individuals may require additional procedures in the uterine cervix to ensure negative margins.

IPD SHARING:
Plan to Share IPD: Undecided